# Reducing Stigma towards Opioid Use Disorder on Interpersonal and Intrapersonal Levels

Manual of Procedures: Intrapersonal Arm

NCT04693416

2/10/2021

| OVERVIEW | 3 |
|----------------------------|----|
| Objectives | 3 |
| Design and Outcomes | 3 |
| Duration | 4 |
| Sample Size and Population | 4 |
| IRB | 4 |
| Award Information | 4 |
| PROJECT ROSTERS | 5 |
| Investigators | 5 |
| Principal Investigator | 5 |
| Co-Investigators | 5 |
| Consultants | 5 |
| Data Safety Officer | 5 |
| Staff | 5 |
| TRAINING PLAN | 6 |
| Pre-Initiation Training | 6 |
| Ongoing Training | 6 |
| ELIGIBILITY CRITERIA | 6 |
| PROCEDURES | 6 |
| Cascade of Events | 6 |
| Baseline | 6 |
| Follow-Up Visit | 7 |
| Recruitment | 7 |
| Consent | 7 |
| Electronic Consent | 8 |
| Intervention | 8 |
| Incentives | 8 |
| Gift Card Distribution | 9 |
| Gift Card Storage | 9 |
| Adverse Events | 9 |
| Retention | 10 |
| MEASURES | 10 |
| Assessment Schedule | 10 |
| CONTACT INFORMATION | 11 |
| DEMOGRAPHICS | 12 |
| SU-SMS | 13 |

| TREATMENT INITIATION | 15 |
|-----------------------------------|----|
| FEEDBACK & TREATMENT SATISFACTION | 15 |
| OTHER DOCUMENTATION | 17 |
| Gift Card Log – Example | 17 |
| Gift Card Receipt | 19 |

#### **PREFACE**

The purpose of this document is to provide a Manual of Operating Procedures (MOP) for the SMART Supplement Project 5a — Intrapersonal Stigma Reduction. The role of the MOP is to facilitate consistency in protocol implementation and data collection across participants and study staff. Use of the MOP increases the likelihood that the results of the study will be scientifically credible and provides reassurance that participant safety and scientific integrity are closely monitored.

#### **OVERVIEW**

# **Objectives**

The goal of this project is to develop and evaluate the efficacy of a stigma reduction intervention that functions at the Intrapersonal (individual) level. Our intervention will address this cost/benefit evaluation among individuals known to face intersecting stigma of alcohol or substance use disorder and African American race, with treatment elements chosen explicitly to increase the value of treatment using salient forms of reward, and to ease perceived costs through explicit services in an effort to encourage the occurrence of the first treatment visit.

# **Design and Outcomes**

This project consists of a pre-post survey, separated by a two-week interval. All elements of our individual intervention are based in Behavioral Economics theory, with the intention of increasing benefits and reducing costs to facilitate individual decision making and reduce subsequent experienced, anticipated, and associative stigma for the individual seeking treatment.

The primary outcome for Project A is reduction in stigma at two weeks post intervention. This will be assessed by using the Substance Use Stigma Mechanisms Scale.

Secondary outcomes include Addiction Treatment visit attendance (e.g., did they attend the visit that was scheduled?) and Feedback and Satisfaction with treatment.

Duration

Participants will be enrolled at baseline (week 0) and will have one follow-up assessment to be

completed two weeks after enrollment.

Sample Size and Population

Approximately 50 participants will be recruited from the Frayser community of Memphis, at the

recruitment site of Legacy of Legends (or associated venue, as dictated by Legacy events).

Participants must identify as having a substance use problem and must not currently be in

treatment. All participants must be over age 18, able to understand consent procedures, reside in

the Frayser community, identify as African American or mixed race, and have access to a

telephone for retention/follow up.

**IRB** 

Project number: 20-07852-XP

The University of Tennessee Health Science Center IRB (FWA00002301) is the reviewing IRB

for this study. Initial approval was received on 02/05/2020.

**Award Information** 

Funding Agency: National Center for Complementary & Integrative Health (NCCIH)

**Award number**: 3R61AT010604-01S1

Grant Title: Behavioral Economics based stigma reduction intervention for low income, African

American individuals with Opioid Use Disorder. (3R61AT010604-01S1).

**Grant Years:** 

10/1/2020 - 9/30/2021

**Supplement Grant Amount: \$201,631** 

**Program Director Clinical Research** 

Peter Murray, PhD

Division of Extramural Research

National Center for Complementary & Integrative Health (NCCIH)

6707 Democracy Boulevard, Suite 401 Bethesda, Maryland 20892-5475

Phone: 301-496-4054 Email: peter.murray@nih.gov

#### **PROJECT ROSTERS**

# **Investigators**

# **Principal Investigator**

#### Karen Derefinko, PhD

University of Tennessee Health Science Center 66 N. Pauline Street, Suite 649
Memphis, TN 38163
901-448-2526
kderefin@uthsc.edu

### **Co-Investigators**

**James G. Murphy, PhD** - University of Memphis, Department of Psychology *jgmurphy@memphis.edu* 

**Fridtjof Thomas, PhD** - UTHSC, Department of Preventive Medicine *fthomas4@uthsc.edu* 

#### **Consultants**

Joseph Palamar, PhD, MPH - New York University Grossman School of Medicine Public Stigma of Substance Use

Joseph.Palamar@nyulangone.org

Charlie Caswell - New York University Grossman School of Medicine Community Integration Consultant legacyoflegendscdc@gmail.com

# **Data Safety Officer**

**Marion Hare, MD** - UTHSC Department of Preventive Medicine <u>mhare@uthsc.edu</u>

#### Staff

Sarah Hand, MPH, CCRP Research Project Manager shand@uthsc.edu

#### **Unjanae Johnson**

Research Coordinator I

#### TRAINING PLAN

# **Pre-Initiation Training**

The Research Coordinator will be trained in data collection, data entry, adverse event collection, incentive distribution, and informed consent procedures by the Project Manager (Hand). Dr. Derefinko will train the coordinator on intervention delivery and fidelity.

# **Ongoing Training**

Data will be monitored throughout the study so that any quality assurance issues can be handled in a timely manner. Any issues with data collection, data entry, informed consent, and incentive distribution will be monitored by Ms. Hand and will be addressed at biweekly staff meetings. Issues regarding study fidelity will be addressed by Dr. Derefinko as needed.

#### **ELIGIBILITY CRITERIA**

Participants must meet the following eligibility criteria to participate in this study:

- Age 18 or older
- Able to understand consent procedures
- Identify as African American or mixed race,
- Access to telephone for retention/follow up
- Self-identified alcohol or substance use disorder (SUD) related issues, and
- Not currently in treatment for SUD.

#### **PROCEDURES**

#### **Cascade of Events**

#### Baseline

- Engage with potential participants to provide information about participation.
- If interested, complete screening for eligibility/exclusionary criteria.
- Complete informed consent.
- After participants have signed the informed consent form, we will collect the remaining baseline data and deliver the intervention.
  - Administer assessments which include contact information, demographics, and SU-SMS (stigma scale)
  - o Deliver intervention
  - Offer to help schedule appointment at CAS (or other clinic)

- Set appointment date/time for 2-week follow-up visit or call.
- Provide a \$20 Kroger gift card as compensation for enrollment.
  - Kroger gift cards will be given via a hard copy gift card following the <u>incentive</u> procedures.
- If the participant schedules a visit and needs transportation support, schedule a Lyft ride
- Provide participant your contact information to ensure that the Lyft ride can be changed as needed (Lyft is scheduled only through us, not the participant).

#### Follow-Up Visit

- At two weeks post baseline:
- Complete follow-up assessments including SU-SMS, attendance at physician visit, and treatment feedback & satisfaction
- Provide the \$20 Kroger gift card upon completion of visit

This is a general script, but can be changed as needed for each situation.

• Kroger gift cards will be given via a hard copy gift card following the <u>incentive</u> procedures.

#### Recruitment

Potential participants who are being referred for potential substance use disorder treatment will be recruited by the Research Coordinator I and Pastor Caswell through Frayser community events, Impact Ministries events, and Legacy of Legends CDC events.

#### **Recruitment Script**

| | 8 | 1 / | 8 | |
|---|---|---|---|---|
| "Hi, _ | ! My nam | e is | and I am part of the i | research staff with the Department of |
| Preve | ntive Medicino | e at the U | Iniversity of Tennesse | e Health Science Center. You're here today |
| becau | se you agreed | to speak | with us about your fe | eelings about drug and alcohol use, and you'r |
| open i | to hearing abo | ut treatm | nent options. We're do | oing a research study where we ask people |
| questi | ons, have a di | scussion, | and then ask a few m | iore questions. |

If you think you might be interested in being in this study, I can ask you a few questions to see if you're eligible, then we can go through a consent form with you to help you decide if you'd like to participate. Are you interested in seeing if you're eligible?

If a person does not wish to participate, we can still provide a handout or information about how to get treatment.

#### **Consent**

The consent of the adult subject will be obtained at the first study visit at baseline after assessing for eligibility but before any identifying data collection begins.

Inviting the subject to read and sign the consent form is not sufficient for securing informed consent. Study staff will go through the consent form with the participant, reviewing all elements of informed consent as stated in 21 CFR 50 § B and will answer all questions regarding the study.

A copy of the informed consent will be given to the subject and the original(s) will be placed in the subjects' research record. An entry documenting informed consent must also be made in the subjects' research record to confirm that informed consent was obtained prior to any study-related procedures and that the subject received a signed copy. The objection of any subject in word or action to the performance of study procedures will be sufficient for their withdrawal or exclusion from the study. Study procedures will not continue until a signed consent form is received.

#### **Electronic Consent**

This project received approval for alteration of consent through the UTHSC IRB. In circumstances where a participant is unable to consent in person due to COVID restrictions, the participant may be consented using DocuSign.

All standard procedures for consent must be followed including the participant being able to view the document while staff reviews with them, having sufficient time to review the document and ask questions, etc.

#### Intervention

The Intrapersonal Stigma Reduction Intervention will address the stigma of addiction, education about addiction, life goals, deciding whether to disclose addiction, and links to services. These modules are covered in an effort to encourage the occurrence of the first treatment visit at the Center for Addiction Science. See Appendix A for the full intervention script.

#### **Data Collection**

Whether in-person or on the phone, research staff will read aloud the items from each measure for the participant to answer. The staff member will record the responses on the paper forms and will later enter the data electronically.

#### **Incentives**

#### Gift Card Distribution

Participants will receive \$20 upon completion of each visit (baseline and follow-up) in the form of a Kroger gift card. The gift cards will be photocopied or scanned onto the gift card receipt. The staff member will take the receipt, gift cards, and a computer back into the room with the participant and check the gift card balance on the Kroger website before distributing. Once the balance is verified, the staff member will fill out the receipt in front of the participant. Both the

research staff and the participant will sign the receipt verifying the information to be true. We will provide a copy of the receipt to the participant.

#### **Gift Card Storage**

Since this project is remote and we will not have ready access to a safe, a minimal number of gift cards should be checked out each week and stored in the locked briefcase with other study documents. Gift cards should only be checked out of the safe when they are ready to be disbursed to a participant. The remaining gift cards will be kept in the safe on the 6th floor of the Pauline Building. The gift card log will be kept in the safe and filled out each time a gift card is moved in or out of the safe.

#### **Adverse Events**

Adverse events (AE's) are defined as any unfavorable medical occurrence in a human subject, including any abnormal sign, symptom, or disease temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.

Serious adverse events (SAE's) are any adverse event temporally associated with the subject's participation in research that meets any of the following criteria:

- Results in death
- <u>Is life-threatening</u> (places the subject at immediate risk of death from the event as it occurred)
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in a persistent or significant disability/incapacity;
- Results in a congenital anomaly
- Any other adverse event that, based upon appropriate medical judgment, may jeopardize
  the subject's health and may require medical or surgical intervention to prevent one of the
  other outcomes listed in this definition

If a participant experiences any adverse event during the course of the study, we will conduct an assessment, complete an Adverse Event form, and follow the adverse event reporting system as required by our IRB and NIH regulations.

All SAE's that are potentially related to the study are to be reported to the Project Coordinator (Sarah Hand) within one working day. The Project Coordinator will review and escalate to the PI via email within 48 hours of initial documentation.

UTHSC's IRB operating procedures regarding AE's can be found here: <a href="https://www.uthsc.edu/research/compliance/irb/researchers/documents/adverse-event-reporting.pdf">https://www.uthsc.edu/research/compliance/irb/researchers/documents/adverse-event-reporting.pdf</a>

#### Retention

It is the job of the research staff to retain all participants in the study in an attempt to have all participants complete their follow up visit. Staff will use various retention efforts to remain in contact with the participants after enrollment. Staff will also send participants an appointment reminder via text the day before their follow up visit (or via phone if preferred by participant).

Participants will have an additional 2 weeks to make up their missed appointment in order to provide us with the data and so they may receive their compensation. The following retention efforts should be made:

- 1. Calling the participant to check in and/or offer another date to reschedule.
- 2. Texting the participant to offer another date.
- 3. Emailing the participant.
- 4. Mailing a letter to the most recent address on file.

The research staff will cycle through these retention efforts during the 2 weeks to ensure they are doing their due diligence to contact the participant. The visit can be completed over-the-phone or in-person.

#### **MEASURES**

#### **Assessment Schedule**

| Measure | Baseline | Follow-Up |
|---|---|---|
| Contact Information | X | |
| Demographics | X | |
| Substance Use Stigma Mechanisms Scale (SU-SMS) | X | X |
| Agreement to set up intake visit at Center for Addiction<br>Science (or other treatment facility) | X | |
| Attendance at intake visit at Center for Addiction Science (or other treatment facility) | | X |

| Feedback & Treatment Satisfa | ction | | X |
|------------------------------|-------|----|---|
| CONTACT INFORMATION | N | | |
| First: | | | |
| Middle: | | | |
| Last: | | | |
| Street: | | | |
| Apt/Suite: | | | |
| City/State/Zip: | | | |
| Email: | | | |
| Primary Phone: | | | |
| Can we leave a voicemail? | Yes | No | |
| Can we send a text? | Yes | No | |
| Secondary Phone: | | | |
| Can we leave a voicemail? | Yes | No | |
| | Yes | No | |

Can we send a text?

| DEMOGRAPHICS | | | | | | | |
|---|---|---|---|---|---|---|---|
| Date of Birth: | | | | | | | |
| Gender: | Male | | Fem | ale | | Transgender | |
| Sex at birth: | Male | | Fem | ale | | | |
| Race (circle all that apply): | African American<br>Black | or | Wh | ite | | A | laskan Native |
| ' | Pacific Islander | | Native A | merican | Ot | ther: _ | |
| Are you of Spanish,<br>Hispanic, or Latino<br>origin? | Ye | S | No | | | ) | |
| | • | | , | | | | |
| Current Marital<br>Status: | Married or living married | g as | W | idowed | | Divorced | |
| ' | Separated | | Single, 1 | never marrie | ed | | |
| Current Household<br>Income per year: | Less than \$10,000 | \$10,0 | 000-19,999 | \$20,000 | \$20,000-29,999 | | \$30,000-39,999 |
| | \$40,000-49,999 | \$50,0 | 000-59,999 | \$60,000 | 0-69,9 | 999 | \$70,000-79,999 |
| | \$80,000-89,999 | \$90,0 | 690,000-99,999 Over \$1 | | 100,0 | 000 | Unsure |
| Highest level of schooling completed: | 8 <sup>th</sup> grade or less | 9 <sup>th</sup> -11 <sup>th</sup> grade | | 11 <sup>th</sup> grade 12 <sup>th</sup> grade o | | GED | Associate's degree |
| ı | Vocational or<br>Trade School | Some | e college | Bachelor's degree | | Graduate degree | |

# **SU-SMS**

How often have people treated you this way in the past because of your alcohol and/or drug use history? Please circle your response.

| | | Never | Not<br>often | Somewhat often | Often | Very<br>Often |
|---|---|---|---|---|---|---|
| 1. | Family members have thought that I cannot be trusted. | 1 | 2 | 3 | 4 | 5 |
| 2. | Family members have looked down on me. | 1 | 2 | 3 | 4 | 5 |
| 3. | Family members have treated me differently. | 1 | 2 | 3 | 4 | 5 |
| 4. | Healthcare workers have not listened to my concerns. | 1 | 2 | 3 | 4 | 5 |
| 5. | Healthcare workers have thought that I'm pill shopping, or trying to con them into giving me prescription medications to get high or sell. | 1 | 2 | 3 | 4 | 5 |
| 6. | Healthcare workers have given me poor care. | 1 | 2 | 3 | 4 | 5 |

How likely is it that people will treat you in the following ways in the future because of your alcohol and/or drug use history?

| Very<br>unlikely | Unlikely | Neither<br>unlikely nor<br>likely | Likely | Very<br>likely |
|---|---|---|---|---|
|---|---|---|---|---|

| 1. | Family members will think that I cannot be trusted. | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|---|
| 2. | Family members will look down on me. | 1 | 2 | 3 | 4 | 5 |
| 3. | Family members will treat me differently. | 1 | 2 | 3 | 4 | 5 |
| 4. | Healthcare workers will not listen to my concerns. | 1 | 2 | 3 | 4 | 5 |
| 5. | Healthcare workers will think that I'm pill shopping, or trying to con them into giving me prescription medications to get high or sell. | 1 | 2 | 3 | 4 | 5 |
| 6. | Healthcare workers will give me poor care. | 1 | 2 | 3 | 4 | 5 |

How do you feel about your alcohol and/or drug use history?

| | | Strongly<br>disagree | Disagree | Neither<br>disagree<br>nor agree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| 1. | Having used alcohol and/or drugs makes me feel like I'm a bad person. | 1 | 2 | 3 | 4 | 5 |
| 2. | I feel I'm not as good as others because I used alcohol and/or drugs. | 1 | 2 | 3 | 4 | 5 |
| 3. | I feel ashamed of having used alcohol and/or drugs. | 1 | 2 | 3 | 4 | 5 |

| 4. | I think less of myself because I used alcohol and/or drugs. | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|---|
| 5. | Having used alcohol and/or drugs makes me feel unclean. | 1 | 2 | 3 | 4 | 5 |
| 6. | Having used alcohol and/or drugs is disgusting to me. | 1 | 2 | 3 | 4 | 5 |

| TREATMENT INITIATION | | |
|---|---|---|
| Did you go to any facility for substance use treatment since we last spoke? | Yes | No |
| If yes, where did you get treatment? | | |

| FE | FEEDBACK & TREATMENT SATISFACTION | | | |
|---|---|---|---|---|
| 1. | How interesting did you find this study? | Totally bad, boring | ок | Excellent, it was great |
| 2. | What made you want to enroll in this study? (select all that apply) | I wanted help getting treatment | Gift cards | Other |
| 3. | How personally relevant did you find this study? | Not at all relevant | Somewhat<br>relevant | Very relevant |
| 4. | How effective do you think this study was in helping you start treatment? | Not at all ettective | Somewhat effective | Very Effective |
| 5. | For those who haven't sought treatment: How likely you are to seek treatment in the near future? | Unlikely | Unsure | Likely |
| 6. | How effective, overall, do you think this program will be in helping substance users seek treatment? | 1 = Not useful or effective | | |
| | | | ve. The best treat | ment I could imagine. |

| | What was the most effective part of this study for you? | (Open ended) |
|---|---|---|
| 8. | Can you think of any ways to make this study more effective and user-friendly? | (Open ended) |

# OTHER DOCUMENTATION

# Gift Card Log – Example

# **Kroger \$20 Gift Cards**

| | -8- | | | |
|---|---|---|---|---|
| Card Number | LOG IN<br>Initials | LOG IN<br>Date | DISPENSE<br>Date | LOG OUT<br>Initials |

| C. C. | | $\mathbf{T}$ | • | - 4 |
|---------|------|--------------|------|-----|
| ( -11ff | Card | ĸ | ecen | nt |
| OIII | Caru | 1 | CCCI | pι |

| Study ID |
|----------|
|----------|

The participant and I, the research staff member, checked the balance of the gift card before distribution. We discussed that the Research Study is not responsible for and will not replace lost or stolen gift cards once the gift card has been disbursed.

| Date | / | | |
|-------------------------|---|--------------|----|
| Staff<br>Initials | | GC<br>Amount | \$ |
| Participant<br>Initials | | Quantity | |